CLINICAL TRIAL: NCT00383409
Title: Multivitamins do Not Improve Radiation Therapy Related Fatigue: Results of a Double-Blind Randomized Cross-Over Trial
Brief Title: Multivitamins do Not Improve Radiation Therapy Related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/2005
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Breast Cancer
Keywords: breast; cancer; fatigue; multivitamins
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Fatigue | interventions — Geritol

INTERVENTIONS:
Drug: multivitamins
Drug: placebo

SUMMARY:
Multivitamins (MVi) are broadly used by cancer patients to improve overall health and energy. Fatigue is a common symptom in cancer patients including those receiving radiation therapy. We conducted a trial of MVi versus placebo in patients with breast cancer (BC) undergoing radiation therapy (Rxt) to evaluate if MVi would affect fatigue and quality of life. We randomized patients at the beginning of Rxt treatment to either placebo or Centrum Silver® (Wyeth-Whitehall laboratory). At the middle of the radiation treatments patients were switched from placebo to MVi and vice versa. Patients answered to the EORTC QLQ C-30 quality of life (QOL) and Chalder Fatigue Questionnaires at the beginning, the time of switching and at the end of Rxt. We found that both groups experienced significant decreases in general and physical fatigue at the end of the course of placebo compared to the assessment prior to this treatment. We also observed significant improvements in functional and symptoms in the patients on placebo. When we compared different groups of patients we also observed significantly lower rates of physical and general fatigue in the patients who had just finished a course of placebo as compared to patients finishing course of MVi. We conclude that MVi do not improve radiation related fatigue, and may in fact have a deleterious effect on fatigue and decrease QOL in patients with BC undergoing Rxt.

DETAILED DESCRIPTION:
Multivitamins (MVi) are broadly used by cancer patients to improve overall health and energy. Fatigue is a common symptom in cancer patients including those receiving radiation therapy. We conducted a double blind randomized cross-over trial of MVi versus placebo in patients with breast cancer (BC) undergoing radiation therapy (Rxt) to evaluate if MVi would affect fatigue and quality of life. We randomized forty patients at the beginning of Rxt treatment to either placebo or Centrum Silver® (Wyeth-Whitehall laboratory). At the middle of the radiation treatments patients were switched from placebo to MVi and vice versa. Patients answered to the EORTC QLQ C-30 quality of life (QOL) and Chalder Fatigue Questionnaires at the beginning, the time of switching and at the end of Rxt. When we analyzed the same group of patients throughout the treatment periods, we found that both groups experienced significant decreases in general (p = 0.009; p = 0.001) and physical fatigue scores (p = 0.031; p = 0.029) at the end of the course of placebo compared to the assessment prior to this treatment. We also observed significant improvements in functional (p = 0.026) and symptoms (p = 0.016) score scales of the QOL questionnaire in the patients on placebo. No significant changes were elicited with the use of MVi. When we compared different groups of patients we also observed significantly lower rates of physical and general fatigue in the patients who had just finished a course of placebo as compared to patients finishing course of MVi (0 vs 25% p = 0.035 for both types of fatigue). We conclude that MVi do not improve radiation related fatigue, and may in fact have a deleterious effect on fatigue and decrease QOL in patients with BC undergoing Rxt. Further studies are needed to confirm our findings.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* breast cancer who were to receive radiation therapy to the breast after a conservative surgery or after mastectomy

Exclusion Criteria:

* previous history of radiation therapy,
* chronic anemia,
* depression
* serious psychiatric disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-03; Study Completion 2006-08

PRIMARY OUTCOMES:
fatigue

SECONDARY OUTCOMES:
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Auro Del Giglio, MD, Study Director — FM-ABC
Locations (1):
- Instituto de Radioterapia do ABC - Av. Portugal, 592 -, Santo André, São Paulo, Brazil